CLINICAL TRIAL: NCT03681522
Title: What is the Most Effective Local Anesthesia for Prostate-stained Ultrasonography-guided Biopsy in PPB and PNB?: A Single Center, Prospective, Randomized, Double Arm Study
Brief Title: A Study on the Pain Control Effect of the Anesthetic Method During Prostate Biopsy: Comparison Between Pelvic Plexus Block and Periprosthetic Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Kang Su Cho, associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2018-0211
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Transrectal Systematic Prostate Biopsy Related Pain
Keywords: local anesthesia; prostate, biopsy; transrectal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic plexus block (Experimental): The injections of 2.5 mL of 2% lidocaine were made to the pelvic neurovascular plexus located at the end of the seminal vesicle under Doppler US guidance on each side
  Interventions: Procedure: Pelvic plexus block
- Periprostatic nerve block (Active Comparator): The injections of 2.5 mL of 2% lidocaine were made to the neurovascular bundles at the junction of the prostate-bladder-seminal vesicle.
  Interventions: Procedure: Periprostatic nerve block

INTERVENTIONS:
Procedure: Pelvic plexus block — Injections of 2.5 mL of 2% lidocaine were made to the pelvic neurovascular plexus located at the end of the seminal vesicle under Doppler US guidance on each side
  Arms: Pelvic plexus block
Procedure: Periprostatic nerve block — Injections of 2.5 mL of 2% lidocaine were made to the neurovascular bundles at the junction of the prostate-bladder-seminal vesicle on each side.
  Arms: Periprostatic nerve block

SUMMARY:
This study assesses differences in the effects of pelvic plexus block and periprostatic nerve block among various anesthetic methods that reduce the pain caused by prostate biopsy.

DETAILED DESCRIPTION:
Recently, various types of local anesthetic methods have been attempted to reduce biopsy-related pain leading to changes in the type of anesthetic agents and site of injection. Of these anesthetics and combinations, pelvic plexus block and periprostatic nerve block seem to be the very effective way to control prostate biopsy-related pain. However, few studies have compared these two methods.

ELIGIBILITY:
Inclusion Criteria:

* abnormal prostate finding on digital rectal examination
* serum PSA level of > 2.5 ng/mL
* Transrectal ultrasonographic abnormal lesion

Exclusion Criteria:

* under 50 years old
* a history of previous TRUS-guided biopsy
* chronic prostatitis/pelvic pain
* neurological conditions (dementia, Parkinson disease, or cerebral infarction)
* bleeding diathesis
* active UTI
* hemorrhoids/anal fissure/anal fistula
* known allergy to lidocaine

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale-1 | day 7~14
  Visual analog scale (0-10) during anesthesia procedure higher values represent a worse outcome.
Visual analog scale-2 | day 7~14
  Visual analog scale (0-10) at insertion of ultrasound probe higher values represent a worse outcome.
Visual analog scale-3 | day 7~14
  Visual analog scale (0-10) during biopsy procedure higher values represent a worse outcome.
Visual analog scale-4 | day 7~14
  Visual analog scale (0-10) at 15 min after the biopsy procedure higher values represent a worse outcome.

SECONDARY OUTCOMES:
Rate of Complication | day 14~28
  Complications after biopsy
Procedure time | day 7~14
  Total time taken for prostate biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Medical College Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided